CLINICAL TRIAL: NCT07336030
Title: Effect of Baduanjin Exercise on Health and Wellbeing for Health Sustainability in Diabetic Patients
Brief Title: Effect of Baduanjin Exercise in Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebatullah Hamdy Mahmoud, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/006072
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus
Keywords: baduanjin exercise; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): baduanjin exercise, diaphragmatic breathing and upper and lower limb stretching exercises
  Interventions: Other: baduanjin exercise
- Control group (Active Comparator): diaphragmatic breathing and upper and lower limb stretching exercises
  Interventions: Other: diaphragmatic breathing exercise and upper and lower limb stretching exercise

INTERVENTIONS:
Other: baduanjin exercise — baduanjin exercise is a type of traditional Chinese exercises that combines exercise and mindful breathing. Baduanjin also called eight section brocades Qigong, the combination of physical movement and intention in these exercises creates enjoyable experiences for both the body and the mind.
  Arms: Experimental group
Other: diaphragmatic breathing exercise and upper and lower limb stretching exercise — diaphragmatic breathing exercise is a breathing exercise which focuses on diaphragm muscle as it is the main respiratory muscle. While upper and lower stretching exercises focuses on flexibility and stretching of major muscle compartments of upper and lower limbs.
  Arms: Control group

SUMMARY:
This study is conducted to assess baduanjin exercise for its ability to reduce cortisol levels in type 2 diabetic patients which in turn contributes to lowering blood glucose levels. the potential improvement in blood sugar levels can positively affect patients' quality of life and improving activities of daily living by reducing complications and dependance on medications , so baduanjin exercise supports the concept of health sustainability and enhancing long term wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both sexes diagnosed with type 2 diabetes.
* Patients with type 2 diabetes for 5-10 years.
* Patients are on oral antihyperglycemic drugs.
* Patients with HbA1c levels between 6.5% and 7%
* Age ranges from 50 to 60 years.
* Patients with BMI from 30-34.9 kg/m2.

Exclusion Criteria:

* patients with cardiac problems e.g. heart failure.
* psychological or mental illness.
* musculoskeletal problems.
* neurological problems.
* liver, kidney, lung diseases.
* autoimmune diseases.
* patients with cognitive diseases.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Diabetes quality of life questionnaire | 12 weeks
  diabetes quality of life questionnaire is used for assessing the patient's current condition and for evaluating improvements in quality of life following interventions.

SECONDARY OUTCOMES:
HbA1C | 12 weeks
  HbA1C is a gold standard in diagnosing diabetes and also it is used for follow up after interventions whether drug or other form of therapeutic interventions as baduanjin exercise.
functional capacity | 12 weeks
  functional capacity using timed up and go (TUG) test. TUG test is performed by the patient as he is asked to stand up from a chair and walk a distance of 3 meters in his normal pace then return to sit down. stop watch is used to calculate the time taken to cover this distance.
Katz index | 12 weeks
  one of the most common instruments in measuring Activities of daily living(ADL) disability is the Katz index of independence in ADL

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt